CLINICAL TRIAL: NCT02008773
Title: A Double-Blind Trial of Adjunctive Valacyclovir to Improve Cognition in Early Phase Schizophrenia
Acronym: VISTA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Stanley Medical Research Institute (Other); Sheppard Pratt Health System (Other); University of Maryland (Other); Centers for Behavioral Health, LLC (Unknown); Laureate Institute for Brain Research, Inc. (Other); University of Kansas Medical Center (Other); University of California, Los Angeles (Other); Yale University (Other); Innovative Clinical Research, Inc. (Industry); University of California Riverside at C.I. Trials, Inc.-Inland Empire (Unknown); Clinical Innovations (Industry)
Responsible Party: Principal Investigator, Alan Breier, Psychiatrist, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1310496490
Record Dates: First submitted 2013-12-07; First posted 2013-12-11 (Estimated); Results first posted 2019-01-30 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Schizophrenia
Keywords: schizophrenia; schizoaffective; schizophreniform; inflammatory markers; HSV1; cognition; early psychosis; valacyclovir
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- valacyclovir (Active Comparator): 3000mg daily oral 16 weeks
  Interventions: Drug: Valacyclovir HCI 500 mg tablets
- placebo (Placebo Comparator): placebo 6 capsules daily oral 16 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Valacyclovir HCI 500 mg tablets — Valacyclovir HCI 500 mg capsules 6/day oral for 16 weeks
  Arms: valacyclovir
Drug: placebo — placebo capsules 6/day oral for 16 weeks
  Other Names: placebo capsules
  Arms: placebo

SUMMARY:
The primary aim of the study is to determine the efficacy of adjunctive valacyclovir, in comparison to placebo, to improve visual (Brief Visuospatial Memory Test) and working (composite score of the Spatial Span and Letter Number Span tests) memory in individuals who are HSV-1 positive and early in the course of schizophrenia.

We hypothesize that individuals who are HSV-1 positive, but not those who are HSV-1 negative, will demonstrate significant valacyclovir efficacy for visual and working memory.

DETAILED DESCRIPTION:
One hundred and seventy-five participants (N=70 HSV-1 seropositive and N=105 HSV-1 seronegative) will be randomized 1:1 to receive adjunctive valacyclovir or adjunctive placebo for a 16 week period. The primary outcome that will be assessed is improvement in changes in visual and working memory scores in HSV-1 positive and negative participants over the course of the study. We will also measure the overall cognitive functioning and the severity of psychiatric symptoms over the course of the study and will evaluate the tolerability and safety of valacyclovir treatment in this population. In addition, we will explore the relationship between changes in the levels of inflammatory markers (HSV2, CMV, EBV, CRP, and Toxoplasmosis) and treatment response over the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 40 years of age at study entry.
* Able to give written informed consent.
* DSM IV-TR Diagnosis of schizophrenia, schizophreniform, or schizoaffective disorder as confirmed by Structured Clinical Interview for DSM-IV-TR (SCID)
* Onset of schizophreniform disorder, schizophrenia, or schizoaffective disorder within the past eight years as defined by first medical records documentation of these conditions
* Outpatient or inpatient.
* Clinical stability as defined by:

  1. CGI-S score of less than or equal to 4 (moderately ill) at randomization AND
  2. Participants must not have experienced an exacerbation of their illness within 4 weeks prior to randomization leading to an intensification of psychiatric care in the opinion of the investigator. Examples of intensification of care include, but are not limited to: inpatient hospitalization, day/partial hospitalization, outpatient crisis management, or psychiatric treatment in an emergency room AND
  3. Antipsychotic treatment stability for at least 4 weeks prior to randomization (no change in antipsychotic dosing, addition of any new antipsychotic medication, or discontinuing an antipsychotic medication)
* Fluent in English.
* Female participants of childbearing potential must test negative for pregnancy at screening visit and agree to use a single, effective, medically acceptable method of birth control for the duration of the study.

Exclusion Criteria:

* Known IQ less than 70 as determined by medical history.
* IV drug use within previous three month prior to study entry.
* Any serious active medical condition that affects brain or cognitive functioning (e.g., epilepsy, serious head injury, brain tumor or other neurological disorder) in the investigator's opinion.
* Known medical history of Human Immunodeficiency Virus (HIV)
* Receipt of valacyclovir or chemically-related medication within 2 weeks prior to randomization.
* History of hypersensitivity to valacyclovir or acyclovir as determined by self-report and medical history.
* DSM-IV diagnosis of substance dependence within 3 months of study entry (with the exception of nicotine or caffeine dependence).
* Participants who have participated in a clinical trial with any pharmacological treatment intervention for which they received study-related medication in the 4 weeks prior to screening AND participants currently receiving treatment (within 1 dosing interval plus 4 weeks) with an investigational depot formulation of an antipsychotic medication.
* Females who are pregnant or planning to become pregnant or breastfeeding or planning to do so during the study period.
* Participants with current acute, serious, or unstable medical conditions, including, but not limited to: inadequately controlled diabetes, asthma, COPD, recent cerebrovascular accidents, acute systemic infection or immunologic disease, unstable cardiovascular disorders, malnutrition, or hepatic or renal disease, renal including renal failure, gastroenterologic, respiratory, endocrinologic, neurologic, hematologic including thrombotic thrombocytopenia purpura/hemolytic uremic syndrome, or infectious diseases
* Participants who require concomitant treatment with any other medication other than those allowed as specified in Attachment 2, or with any other medication specifically excluded in Attachment 2.
* Clinically significant electrocardiogram (ECG) abnormality prior to randomization as defined by: participants with a corrected QT interval (Bazett's; QTcB) >450 msec (male) or >470 msec (female) prior to randomization. Repeat ECGs will be conducted at the discretion of the principal investigator or medical designee.
* Test positive for (1) Hepatitis C virus antibody, (2) Hepatitis B surface antigen (HBsAg) with or without positive Hepatitis B core total antibody.
* Participants with moderate to severe renal impairment as defined by creatinine clearance (CrCl) < 60 ml/min (measured by the Cockcroft-Gault equation) at screening.
* Participants with hepatic impairment as defined by liver transaminases or total bilirubin > 3 × upper limit of normal (ULN).
* Participants considered a high risk for suicidal acts - active suicidal ideation as determined by clinical interview OR any suicide attempt in 90 days prior to screening.
* Participants who demonstrate overtly aggressive behavior or who are deemed to pose a homicidal risk in the investigator's opinion.
* Participants currently receiving cognitive remediation therapy at time of study entry
* Participants who have had electroconvulsive therapy (ECT) within 12 months of study entry or who will have ECT at any time during the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 170 (Actual)
Dates: Start 2014-03-26 (Actual); Primary Completion 2017-06-20 (Actual); Study Completion 2017-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Breier, MD, Principal Investigator — Indiana University; Faith Dickerson, PhD, Principal Investigator — Shepard Pratt Health System; Robert Buchanan, MD, Principal Investigator — University of Maryland; Robert Litman, MD, Principal Investigator — Centers for Behavioral Health, LLC; Sheldon Preskorn, MD, Principal Investigator — University of Kansas (KUMC); Brent Wurfel, MD, PhD, Principal Investigator — Laureate Institute for Brain Research; Stephen Marder, MD, Principal Investigator — University of California, Los Angeles; Keith Nuechterlein, PhD, Principal Investigator — University of California, Los Angeles; Deepak D'Souza, MD, Principal Investigator — Yale University; Rishi Kakar, MD, Principal Investigator — Innovative Clinical Research, Inc.; Gerald Maguire, MD, Principal Investigator — University of California, Riverside; Diane Highum, MD, Principal Investigator — Clinical Innovations; Evagelos Coskinas, MD, PhD, Principal Investigator — Clinical Innovations
Locations (13):
- United States (13):
  - C.I. Trials, Inc.-Los Angeles County, Bellflower, California
  - University of California, Los Angeles, Los Angeles, California
  - University of California, Riverside at C.I. Trials, Inc.-Inland Empire, Riverside, California
  - C.I. Trials, Inc.-Orange County, Santa Ana, California
  - Yale University, New Haven, Connecticut
  - Innovative Clinical Research, Inc., Lauderhill, Florida
  - Prevention and Recovery Center for Early Psychosis, Indianapolis, Indiana
  - Indiana University Psychotic Disorders Clinic, Indianapolis, Indiana
  - University of Kansas Medical Center-Witchita, Wichita, Kansas
  - Maryland Psychiatric Research Center, Baltimore, Maryland
  - Centers for Behavioral Health, LLC, Rockville, Maryland
  - Sheppard Pratt Health System, Towson, Maryland
  - Laureate Institute for Brain Research, Tulsa, Oklahoma

REFERENCES:
- [Derived] Breier A, Buchanan RW, D'Souza D, Nuechterlein K, Marder S, Dunn W, Preskorn S, Macaluso M, Wurfel B, Maguire G, Kakar R, Highum D, Hoffmeyer D, Coskinas E, Litman R, Vohs JL, Radnovich A, Francis MM, Metzler E, Visco A, Mehdiyoun N, Yang Z, Zhang Y, Yolken RH, Dickerson FB. Herpes simplex virus 1 infection and valacyclovir treatment in schizophrenia: Results from the VISTA study. Schizophr Res. 2019 Apr;206:291-299. doi: 10.1016/j.schres.2018.11.002. Epub 2018 Nov 23. PMID 30478008
- See also: Centers for Behavioral Health, LLC — http://www.cbhhealth.com/
- See also: Laureate Institute for Brain Research — http://www.laureateinstitute.org/
- See also: Kansas University School of Medicine, Psychiatry — http://wichita.kumc.edu/psychiatry-and-behavioral-sciences.html

RESULTS

PARTICIPANT FLOW:
Groups:
- HSV1+ Placebo: HSV1 positive subjects assigned to the HSV1+ placebo arm
- HSV1+ Valacyclovir: HSV1 positive subjects assigned to the Valacyclovir study treatment arm
- HSV1- Placebo: HSV1 negative subjects assigned to the placebo arm
- HSV1- Valacyclovir: HSV1 negative subjects assigned to the Valacyclovir study treatment arm
Period: Overall Study
Arm/Group | HSV1+ Placebo | HSV1+ Valacyclovir | HSV1- Placebo | HSV1- Valacyclovir
Started | 40 | 34 | 46 | 50
Completed | 27 | 25 | 32 | 38
Not Completed | 13 | 9 | 14 | 12
Not completed — Adverse Event | 3 | 3 | 1 | 2
Not completed — Medication Non-compliance | 2 | 1 | 3 | 2
Not completed — Withdrawal by Subject | 8 | 4 | 7 | 6
Not completed — Lost to Follow-up | 0 | 1 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HSV1+ Placebo | HSV1+ Valacyclovir | HSV1- Placebo | HSV1- Valacyclovir | Total
Number analyzed (Participants) | 40 | 34 | 46 | 50 | 170
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 40 | 34 | 46 | 50 | 170
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (6.2) | 29.9 (6.1) | 25.3 (4.9) | 27.4 (6.0) | 28.15 (2.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 4 | 12 | 44
  Male | 26 | 20 | 42 | 38 | 126
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 20 | 23 | 23 | 29 | 95
  White | 12 | 7 | 18 | 4 | 41
  More than one race | 8 | 4 | 5 | 17 | 34
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 40 | 34 | 46 | 50 | 170

OUTCOME MEASURES:

1. Primary Outcome: Visual Memory
Description: To determine the efficacy of adjunctive valacyclovir, in comparison to placebo, to improve visual memory (Brief Visuospatial Memory Test) in individuals who are HSV-1 positive and early in the course of schizophrenia. The Brief Visuospatial Memory Test is a subscale of the MATRICS Consensus Cognitive Battery (MCCB) and was used to assess visual memory.
  The BVMT consists of three trials in which participants must recall shapes by drawing figures on a blank page after being given the opportunity to memorize the figures for 10 seconds. Each page consists of six figures. Points are awarded based on the accuracy of the drawn figure and by correct placement on the page. A minimum of 0 to 12 points are awarded per trial, so a participant can score between 0 and 36 points for all three trials. The raw score is then converted to a t-score, normed by age and sex. The min and max t-scores are between 0-100, a higher t-score representing a better outcome.
Time Frame: Baseline, 8 weeks, and 16 weeks
Measure: Least Squares Mean (Standard Error); unit: visual memory scores
Arm/Group | HSV1+ Valacyclovir | HSV1+ Placebo | HSV1- Valacyclovir | HSV1- Placebo
Number analyzed (Participants) | 34 | 40 | 50 | 46
visual memory scores
  MATRICS Brief Visuospatial Memory Baseline | 37.1 (2.1) | 33.9 (1.9) | 39.6 (1.7) | 34.2 (1.9)
  MATRICS Brief Visuospatial Memory Week 8 | 38.2 (2.1) | 34.6 (1.9) | 39.4 (1.7) | 38.0 (1.9)
  MATRICS Brief Visuospatial Memory Week 16 | 39.6 (2.1) | 37.3 (1.9) | 42.2 (1.7) | 41.3 (1.9)

2. Primary Outcome: Working Memory
Description: Determine the efficacy of adjunctive valacyclovir, in comparison to placebo, on working memory (composite score of the Wechsler Memory Scale-III: Spatial Span and Letter Number Span tests). WMS has 2 sections in which a subject recalls increasingly difficult sequences. The total raw score range for both sections is 0-32. The raw score is then converted to a tscore based on normative ranges by age and sex, ranging from 0-100. For both the raw and tscore a higher score reflects better performance.
  LNS consists of 24 increasingly difficult sequences of letters and numbers that a subject is to recall and repeat back in Numeric-Alpha sequential order. The total raw score range is 0-24. The raw score is then converted to a tscore based on normative ranges by age and sex, ranging from 0-100. For both the raw and tscore a higher score reflects better performance. The Working Memory composite score is calculated by summing the WMS and LNS tscores, a higher tscore reflects better performance.
Time Frame: Baseline, 8 weeks, and 16 weeks
Measure: Least Squares Mean (Standard Error); unit: Working Memory Scores
Arm/Group | HSV1+ Valacyclovir | HSV1+ Placebo | HSV1- Valacyclovir | HSV1- Placebo
Number analyzed (Participants) | 34 | 40 | 50 | 46
Working Memory Scores
  MATRICS Working Memory Scores at Baseline | 31.8 (1.9) | 34.1 (1.8) | 40.7 (1.6) | 35.5 (1.8)
  MATRICS Working Memory Scores at 8 weeks | 34.4 (1.9) | 34.7 (1.8) | 41.6 (1.6) | 39.5 (1.8)
  MATRICS Working Memory Scores at 16 weeks | 34.7 (1.9) | 36.4 (1.8) | 42.6 (1.6) | 39.0 (1.8)

3. Secondary Outcome: Cognitive Performance
Description: To evaluate the efficacy of adjunctive valacyclovir, in comparison to placebo, to improve general cognitive performance as measured by the MATRICS Consensus Cognitive Battery composite score in HSV1 + and - participants. MCCB is comprised of 10 tests, Trail Making Test Part A; Brief Assessment in Cognition in Schizophrenia Symbol Coding; Hopkins Verbal Learning Test-Revised; Wechsler Memory Scale-III Spatial Span; Letter Number Sequencing; Neuropsychological Assessment Battery Mazes; Brief Visuospatial Memory Test-Revised; Category Fluency Animal Naming; Mayer-Salovey-Caruso Emotional Intelligence Test Managing Emotions; and Continuous Performance Test-Identical Pairs. For each test, a score is derived based on the raw item values. Each of the individual item raw scores is standardized to age and gender corrected tscores which are then summed to convert into a composite score ranging from <214->486 based on the MCCB scoring manual, with a higher score reflecting better performance.
Time Frame: Baseline, 8 Weeks, and 16 weeks
Measure: Least Squares Mean (Standard Error); unit: MATRICS Composite Scores
Arm/Group | HSV1+ Valacyclovir | HSV1+ Placebo | HSV1- Valacyclovir | HSV1- Placebo
Number analyzed (Participants) | 34 | 40 | 50 | 46
MATRICS Composite Scores
  MATRICS Overall Composite Score at baseline | 27.8 (2.3) | 29.4 (2.1) | 34.8 (1.9) | 30.2 (2.2)
  MATRICS Overall Composite Score at 8 weeks | 27.8 (2.3) | 30.0 (2.1) | 35.6 (1.9) | 33.3 (2.2)
  MATRICS Overall Composite Score at 16 weeks | 29.6 (32.6) | 32.6 (2.1) | 39.2 (1.9) | 36.4 (2.2)

4. Secondary Outcome: Functional Performance
Description: To evaluate the efficacy of adj. valacyclovir to improve functional performance and quality of life (QOL) as measured by the UCSD Performance-Based Skills Assessment, Version B (UPSA-B); QOL Enjoyment and Satisfaction Questionnaire Short Form (Q-LES); and Personal and Social Performance Scale (PSP). The UPSA-B is a performance-based assessment of improvement in functional capacity.Participants are asked to role-play communication and finance tasks. Scores are assigned for each of the 2 subscales and formula is used to calculate a total score (0-100). A higher score reflects better performance. The Q-LES, 16 item scale yields a raw total score, ranging from 14-70, with a higher score representing higher QOL. The PSP scale is a single item scale assessing 4 domains of functioning: personal&social relationships, socially useful activities, self-care, and disturbing&aggressive behaviors. An adjusted score from 0-100 is generated, a higher score reflects better functioning.
Time Frame: Baseline, 8 weeks, and 16 weeks
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | HSV1+ Valacyclovir | HSV1+ Placebo | HSV1- Valacyclovir | HSV1- Placebo
Number analyzed (Participants) | 34 | 40 | 50 | 46
Scores on a Scale
  UPSA-B Total Score at Baseline | 72.6 (2.5) | 71.8 (2.4) | 71.9 (2.2) | 73.4 (2.4)
  UPSA-B Total Score at 8 weeks | 73.4 (2.5) | 74.5 (2.4) | 75.3 (2.2) | 78.6 (2.4)
  UPSA-B Total Score at 16 weeks | 76.7 (2.5) | 75.6 (2.4) | 77.5 (2.2) | 78.8 (2.4)
  Q-LES-Q-SF Total Score at Baseline | 47.8 (1.6) | 50.8 (1.5) | 53.0 (1.3) | 49.4 (1.5)
  Q-LES-Q-SF Total Score at 8 weeks | 50.9 (1.6) | 51.4 (1.5) | 52.6 (1.3) | 50.7 (1.5)
  Q-LES-Q-SF Total Score at 16 weeks | 49.3 (1.6) | 53.7 (1.5) | 54.0 (1.3) | 52.7 (1.5)
  PSP Adjusted Score at Baseline | 55.4 (2.1) | 58.2 (2.0) | 59.9 (1.8) | 59.2 (2.0)
  PSP Adjusted Score at 8 weeks | 55.6 (2.1) | 60.5 (2.0) | 61.7 (1.8) | 61.4 (2.0)
  PSP Adjusted Score at 16 weeks | 58.3 (2.1) | 60.8 (2.0) | 61.3 (1.8) | 61.5 (2.0)

5. Secondary Outcome: Psychosis Symptoms
Description: To evaluate the efficacy of adj. valacyclovir for general and positive symptoms (sxs) as measured by the PANSS total and factor scores and negative sxs as measured by the NSA-16.The PANSS contains 30 items that assess sxs of psychotic d/os.Positive sxs are rated on 7 items, negative sxs on 7 items, and general psych. on 16 items.Scores for each item range from 1-7.Positive total scores ranging from 7-49, negative total scores ranging from 7-49, and general psych. scores ranging from 16-112.Total scores for all items range from 30-210.Additionally a factor score can be derived for Cognition/Disorganization by using scores from 7 items and ranges from 7-49.For factor and total scores a lower score reflects fewer sxs.The NSA-16 is used to rate behaviors commonly associated with negative sxs of schizophrenia.The scale rates subjects on 16 anchors from 1 to 6.The total score is the sum of the 16 specific items and ranges from 16 to 96; a higher score indicates greater severity of illness.
Time Frame: Baseline, 4 weeks, 8 weeks, 12 weeks, and 16 weeks
Measure: Least Squares Mean (Standard Error); unit: Symptom Scale Scores
Arm/Group | HSV1+ Valacyclovir | HSV1+ Placebo | HSV1- Valacyclovir | HSV1- Placebo
Number analyzed (Participants) | 34 | 40 | 50 | 46
Symptom Scale Scores
  PANSS Total Score at Baseline | 66.4 (2.7) | 61.1 (2.5) | 58.9 (2.3) | 64.2 (2.6)
  PANSS Total Score at 4 weeks | 64.8 (2.7) | 60.5 (2.5) | 58.0 (2.3) | 62.1 (2.6)
  PANSS Total Score at 8 weeks | 64.0 (2.7) | 59.5 (2.5) | 57.3 (2.3) | 63.5 (2.6)
  PANSS Total Score at 12 weeks | 62.6 (2.7) | 59.3 (2.5) | 56.0 (2.3) | 61.1 (2.6)
  PANSS Total Score at 16 weeks | 65.1 (2.7) | 57.9 (2.5) | 56.0 (2.3) | 58.9 (2.6)
  PANSS Positive Symptom Factor Score at Baseline | 20.5 (1.0) | 19.3 (10) | 17.2 (0.9) | 19.3 (1.0)
  PANSS Positive Symptom Factor Score at 4 weeks | 20.7 (1.0) | 18.8 (1.0) | 17.1 (0.9) | 18.7 (1.0)
  PANSS Positive Symptom Factor Score at 8 weeks | 20.1 (1.0) | 18.4 (1.0) | 16.8 (0.9) | 18.7 (1.0)
  PANSS Positive Symptom Factor Score at 12 weeks | 19.2 (1.0) | 18.0 (1.0) | 16.0 (0.9) | 18.3 (1.0)
  PANSS Positive Symptom Factor Score at 16 weeks | 19.1 (1.0) | 17.1 (1.0) | 16.1 (0.9) | 17.2 (1.0)
  PANSS Negative Symptom Factor Score at Baseline | 17.1 (1.1) | 14.2 (1.0) | 15.6 (0.9) | 16.0 (1.0)
  PANSS Negative Symptom Factor Score at 4 weeks | 16.8 (1.1) | 15.0 (1.0) | 15.4 (0.9) | 15.5 (1.0)
  PANSS Negative Symptom Factor Score at 8 weeks | 16.5 (1.1) | 15.3 (1.0) | 14.9 (0.9) | 16.0 (1.0)
  PANSS Negative Symptom Factor Score at 12 weeks | 16.6 (1.1) | 14.7 (1.0) | 14.7 (1.0) | 16.0 (1.0)
  PANSS Negative Symptom Factor Score at 16 weeks | 17.5 (1.1) | 14.8 (1.0) | 14.8 (1.0) | 14.8 (1.0)
  PANSS Cognitive/Disorganized Factor Score at Base | 13.7 (0.7) | 13.5 (0.6) | 12.5 (0.6) | 13.2 (0.6)
  PANSS Cognitive/Disorganized Factor Score at 4 wks | 14.0 (0.7) | 12.7 (0.6) | 12.3 (0.6) | 13.0 (0.6)
  PANSS Cognitive/Disorganized Factor Score at 8 wks | 14.0 (0.7) | 12.8 (0.6) | 11.9 (0.6) | 13.7 (0.6)
  PANSS Cognitive/Disorganized Factor Score at 12 wk | 13.6 (0.7) | 12.7 (0.6) | 12.2 (0.6) | 13.0 (0.6)
  PANSS Cognitive/Disorganized Factor Score at 16 wk | 14.6 (0.7) | 12.5 (0.6) | 12.1 (0.6) | 12.4 (0.6)
  NSA-16 Total Score at Baseline | 44.5 (2.3) | 40.2 (2.2) | 42.5 (2.0) | 41.7 (2.2)
  NSA-16 Total Score at 4 weeks | 43.3 (2.3) | 40.2 (2.2) | 42.7 (2.0) | 41.1 (2.2)
  NSA-16 Total Score at 8 weeks | 44.4 (2.3) | 39.9 (2.2) | 41.5 (2.0) | 41.5 (2.2)
  NSA-16 Total Score at 12 weeks | 43.7 (2.3) | 40.6 (2.2) | 41.0 (2.0) | 42.1 (2.2)
  NSA-16 Total Score at 16 weeks | 46.5 (2.3) | 39.9 (2.2) | 41.5 (2.0) | 41.1 (2.2)

6. Secondary Outcome: Functional Performance
Description: To evaluate the efficacy of adjunctive valacyclovir, compared to placebo, to improve to improve global functional assessments as measured by the Clinical Global Impressions Severity Scale (CGI-S). The CGI-S is a single 7-point Likert scale rating severity of psychopathology on a scale of 1 (normal, not ill) to 7 (very severely ill).
Time Frame: Baseline, 8 weeks, and 16 weeks
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | HSV1+ Valacyclovir | HSV1+ Placebo | HSV1- Valacyclovir | HSV1- Placebo
Number analyzed (Participants) | 34 | 40 | 50 | 46
scores on a scale
  CGI-S Scores at Baseline | 3.6 (0.1) | 3.6 (0.1) | 3.5 (0.1) | 3.6 (0.1)
  CGI-S Scores at 4 weeks | 3.6 (0.1) | 3.5 (0.1) | 3.5 (0.1) | 3.5 (0.1)
  CGI-S Scores at 8 weeks | 3.5 (0.1) | 3.3 (0.1) | 3.4 (0.1) | 3.5 (0.1)
  CGI-S Scores at 12 weeks | 3.5 (0.1) | 3.5 (0.1) | 3.4 (0.1) | 3.5 (0.1)
  CGI-S Scores at 16 weeks | 3.5 (0.1) | 3.4 (0.1) | 3.3 (0.1) | 3.5 (0.1)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout the course of subject participation in the 16 week study.
Arm/Group | Valacyclovir | Placebo
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/86
Serious Adverse Events (participants affected / at risk) | 3/84 | 4/86
Other Adverse Events (participants affected / at risk) | 5/84 | 0/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Valacyclovir (N=84) | Placebo (N=86)
Psychotic Illness Exacerbation (Psychiatric disorders) | 3 (3) | 4 (7)
Diabetic Ketoacidosis (Endocrine disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Valacyclovir (N=84) | Placebo (N=86)
Nausea (Gastrointestinal disorders) | 5 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-08): https://cdn.clinicaltrials.gov/large-docs/73/NCT02008773/Prot_SAP_000.pdf